CLINICAL TRIAL: NCT05770323
Title: The Association Between Serum Uric Acid Level and Acute Coronary Syndrome in_hospital Outcomes
Brief Title: Association Between Uric Acid and Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadeer Hassan Abdelaty, Resident doctor at sohag University, Sohag University
Other Study IDs: Uric acid in ACSs
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with normal uric acid levels: Patient with uric acid level (2.5_6)for femal and (3_7)for males
  Interventions: Diagnostic Test: Uric acid level
- Patients with elevated uric acid level (hyperurecemia): Uric acid level more than 7 for males and more than 6 for female
  Interventions: Diagnostic Test: Uric acid level

INTERVENTIONS:
Diagnostic Test: Uric acid level — Uric acid will be measured for all Patients with acute coronary syndrome and result will be analysed

SUMMARY:
The aim of the study is to acess the association between admission serum uric acid level and in_hospital outcomes in patients with acute coronary syndromes

DETAILED DESCRIPTION:
Prospective study

1. To acess patients with acute coronary syndrome including one of (typical Chest pain _ECGchanges _elevated cardic enzyme)
2. the complication occur in patients with hyperurecemia and those with normal uric acid

ELIGIBILITY:
Inclusion Criteria:

all patients with acute coronary syndrome with one of the Following

* Typical Chest pain
* ECG changes
* Elevated cardiac enzyme

Exclusion Criteria:

* patients aged less than 18 years
* patients with gout
* patients with treated with diuretics
* Patient with CKD
* Patient with chronic haemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Patient admited to sohag University in CCU with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-22 (Estimated); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Association between serum uric acid level and acute coronary syndrome in hospital outcomes | From the day of admission and 30 days post discharge
  Comparision between Patient with hyperurecemia and those with normal uric acid level

REFERENCES:
- [Background] Maloberti A, Biolcati M, Ruzzenenti G, Giani V, Leidi F, Monticelli M, Algeri M, Scarpellini S, Nava S, Soriano F, Oreglia J, Sacco A, Morici N, Oliva F, Piani F, Borghi C, Giannattasio C. The Role of Uric Acid in Acute and Chronic Coronary Syndromes. J Clin Med. 2021 Oct 16;10(20):4750. doi: 10.3390/jcm10204750. PMID 34682873